CLINICAL TRIAL: NCT04193397
Title: Effects of Physical Training on Physical and Functional Fitness, Physical Activity Level, Endothelial Function, Hemodynamic Variables, Bone Metabolism and Quality of Life of Post-bariatric Patients: a Randomized Controlled Trial
Brief Title: Effects of Physical Training on Health Markers of Post-bariatric Patients
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BARexe
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery
Keywords: Obesity; Muscle mass; Muscle strength; Bone mineral density; Bone microarchitecture
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention group will perform a supervised resistance training program, while non-exercised control group will receive the standard clinical follow-up and shall not change their physical activity behavior (Study 1) and Post-bariatric group or non-bariatric control group (Study 2)
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Post-bariatric patients - Intervention group
  Interventions: Behavioral: Exercise training
- No intervention (No Intervention): Post-bariatric patients - Non-exercised control group

INTERVENTIONS:
Behavioral: Exercise training — Resistance training program performed during 6 months, 3 sessions per week
  Arms: Exercise training

SUMMARY:
The purpose of this clinical trial is to study the effects of resistance training program on physical-functional fitness, muscle mass and strength, endothelial function, blood pressure, biochemical markers of cardiovascular risk and bone metabolism, density and microstructure and quality of life of post-bariatric patients (Study 1). To compare the bone and muscle changes in post-bariatric patients by Roux-en-Y Gastric Bypass Surgery with non-bariatric controls, as well as to correlate these health indicators with surgery time and weight loss (Study 2).

DETAILED DESCRIPTION:
Randomized controlled trial (Study 1) will feature post-bariatric patients in outpatient care at the public health unit. The post-bariatric patients will be randomized through a random code generator software (www.randomization.com) at a ratio of 1:1, into two groups: a) Intervention group - that will perform a supervised RT program for 6-months or b) Non-exercised control group - that will receive the standard clinical follow-up and shall not change their physical activity behavior. The exercise sessions will include: a) 10-min specific warm-up, consisting of one set of 20 repetitions with loads corresponding to 50% of the resistance used in the first exercise of the training session; b) 45-min of resistance exercises for the upper and lower body (8 single and multi-joint exercises with free weights and machines, including seated rowing, leg press, bench press, leg flexion, pull down, leg extension, shoulder press, and abdominal exercises), performed with 2-3 sets of 8 to 12 repetitions with loads ≥ 70% of one-repetition maximum (1RM) interspersed with 2 min intervals between sets; c) 5-min recovery with stretch and cool-down exercises. During six months, all training sessions will occur three times a week on nonconsecutive days. The outcomes will be assessed by dual energy X-ray emission densitometry (DXA); high resolution peripheral quantitative computed tomography (HR-pQCT), repetition maximum, handgrip strength; biochemical analysis (blood lipid profile, blood glucose and biomarkers of bone formation and absorption and calcium metabolism); venous occlusion plethysmography and nailfold videocapillaroscopy; blood pressure measurement and 36-Item Short-form Health Survey. The cross-sectional study (Study 2) will have 2 groups: post-bariatric patients group (BG) and control group (CG) - non-bariatric controls. Outcomes will be assessed by DXA; HR-pQCT; handgrip strength and biochemical analysis (blood lipid profile, blood glucose and biomarkers of bone formation and absorption and calcium metabolism).

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to Roux-en-Y gastric bypass
* Aging 18 to 50-years
* At least 12 months from surgery

Exclusion criteria:

* Smoking
* Alcoholism
* Gestation
* Cardiovascular disease
* Respiratory disease
* Neurological disease
* Infectious disease
* Endocrine disease
* Musculoskeletal impairments
* Use of hormonal replacement therapy that influence bone metabolism
* Use of medications that influence bone metabolism
* Start some physical exercise program during the study
* Excess weight loss <50%
* Use drugs that interfere with weight
* Revisional bariatric surgery
* Regular physical exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline body composition at 6 months | Baseline and 6 months of follow-up
  Muscle mass and body mineral density will be assessed by Dual-energy X-ray Absortiometry
Changes from baseline bone microarchitecture at 6 months | Baseline and 6 months of follow-up
  Bone microarchitecture will be assessed by High-resolution peripheral quantitative computed tomography
Changes from baseline muscle strength at 6 months | Baseline and 6 months of follow-up
  Muscle strength will be evaluated by one repetition maximum test and handgrip strength
Changes from baseline blood biomarkers at 6 months | Baseline and 6 months of follow-up
  Bone formation and reabsorption biomarkers will be evaluated by blood sample collection
Changes from baseline blood biomarkers at 6 months | Baseline and 6 months of follow-up
  Metabolic profile will be evaluated by blood sample collection

SECONDARY OUTCOMES:
Changes from baseline quality of life indicators at 6 months | Baseline and 6 months of follow-up
  Quality of life indicators will be evaluated by 36-Item Short-form Health Survey
Changes from baseline cardiovascular risk factors at 6 months | Baseline and 6 months of follow-up
  Cardiovascular risk factors will be evaluated by body mass index, waist circumference, blood pressure, triglycerides, HDL-c, LDL-c, total cholesterol, and fasting glycemia
Changes from baseline anthropometric markers at 6 months | Baseline and 6 months of follow-up
  Anthropometric markers will be determined by a digital scale and wall-mounted stadiometer
Changes from baseline hemodynamic measurement at 6 months | Baseline and 6 months of follow-up
  Blood pressure and heart rate will be assessed by a digital sphygmomanometer
Changes from baseline endothelial function at 6 months | Baseline and 6 months of follow-up
  Endothelial function will be evaluated by venous occlusion plethysmography and periungual videocapilaroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Guilherme K De Aguiar, PhD, Principal Investigator — Rio de Janeiro State University, Rio de Janeiro, RJ, Brazil
Locations (1):
- Laboratory for Clinical and Experimental Research on Vascular Biology, Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes KG, das Gracas Coelho de Souza M, da Costa Tavares Bezerra M, Bessa LM, Farinatti P, Bouskela E, Madeira M, Kraemer-Aguiar LG. Effects of physical training on physical and functional fitness, physical activity level, endothelial function, hemodynamic variables, bone metabolism, and quality of life of post-bariatric patients: study protocol for a randomized controlled trial. Trials. 2022 Sep 2;23(1):733. doi: 10.1186/s13063-022-06677-z. PMID 36056396
- [Derived] Lopes KG, Romagna EC, da Silva DS, da Costa Tavares Bezerra M, Leal PRF, da Silva Soares Pinto JE, Bouskela E, das Gracas Coelho de Souza M, Kraemer-Aguiar LG. Metabolic and Inflammatory Profiles of Post-Bariatric Patients with Weight Recidivism. Obes Surg. 2022 Jun;32(6):1849-1855. doi: 10.1007/s11695-022-06025-9. Epub 2022 Mar 23. PMID 35320489